CLINICAL TRIAL: NCT05154942
Title: Acupuncture Combined With DOXO as a Whole Body Probe for Vmax Detection of CYP1A in Vivo
Brief Title: Vmax Detection of Acupuncture-doxofylline as a Whole Probe of CYP1A in Vivo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Collaborators: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20211129
Record Dates: First submitted 2021-11-30; First posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Acupuncture; Drug Interaction
Keywords: Doxofylline; Acupuncture and drug combined technology; Vmax detection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DOXO+electroacupuncture (Experimental): EA is given every day for the first three days before DOXO pumping, and EA is given when DOXO is pumped for 30 minutes each time
  Interventions: Device: DOXO+electroacupuncture
- Non-electroacupuncture (No Intervention): Compared to the experimental group without EA treatment

INTERVENTIONS:
Device: DOXO+electroacupuncture — DOXO+electroacupuncture
  Arms: DOXO+electroacupuncture

SUMMARY:
Preliminary studies have shown that before giving combined acupuncture and medicine anesthesia, electroacupuncture (EA) needs to be started three days before in order to produce a sequential effect. In combined acupuncture and drug anesthesia, the core goal is to use acupuncture to reduce the insufficiency of anesthetics in terms of analgesia, sedation, stable circulation, and protection of organs. However, the mechanism of action behind this combination has not yet been changed. The pharmacodynamics or pharmacokinetics has been convincingly explained, or the degree of recognition is not high, such as whether acupuncture has a specific target in the body, if there is a specific target, where the effect target is located ? Will it affect the metabolic enzymes and will it further affect the efficacy or toxicity of the drugs metabolized by the metabolic enzymes? What effect will it have on the pharmacokinetic mechanism? Given that it may involve complex pharmacodynamics and pharmacokinetic mechanisms, this study will first use doxofylline (DOXO) as a probe to study and explain its effect on metabolic enzymes to further clarify whether it will produce therapeutic drugs Influence.

Doxofylline (DOXO), as an old drug that has been used for many years, has extremely high safety and strong selectivity. It is a clinical drug with an injectable dosage form. Studies have proved that DOXO can be used as a high-quality P450 mixed-function oxidase CYP1A in vivo probe. DOXO is a metabolic clearance-leading drug in the human body, and it must undergo the initiation metabolism of CYP1A in the cell to be transformed into theophylline acetaldehyde ( TA), and then theophylline acetic acid (TAA) and hydroxyethyl theophylline (ETO) produced by disproportionation. Therefore, quantitative detection of TAA and ETO can calculate the maximum activity of CYP1A.

In order to study the kinetics of DOXO and reduce the inconvenience of excessive blood sampling points for long-term continuous administration, we will explore the method of detecting DOXO kinetics by the Vmax method through clinical research to characterize whether acupuncture affects the metabolic enzyme CYP1A

DETAILED DESCRIPTION:
In the face of complex medical challenges, diversified medications, combination medications, compound medications, and precision medications have shown a clear upward trend. Quantitative monitoring of drugs in the body has gradually become a routine. However, this conventional method not only has a lag in time, but also has a scientific principle. There are also serious defects in nature. Time lag is manifested as a lack of predictability and individual differences over time. In principle, drug changes are the result of the body's reaction to drugs.Therefore, the body characteristics related to drug metabolism need to be evaluated first.

The current therapeutic drug monitoring is almost lack of theoretical support. From the perspective of safety and mechanism-based pharmacokinetics, its specific manifestations are as follows: 1. Considering the individual safety, although there is the information support of group medicine, the drug dose must also be tested from a small dose; 2. The plasma drug concentration must be completed by multi-point continuous overall kinetic process test or obtained by model derivation, such as in vitro derivation based on enzymatic Michaelis kinetic parameters; 3. Single point plasma concentration can not replace the overall kinetic model. If necessary, there must be many assumptions and conditions. Therefore, the steady-state single point therapeutic drug monitoring (TDM) test obviously does not have the above three functions. Its data is unreasonably amplified to guide the accurate clinical administration, which will inevitably lead to many defects existing in principle, that is, "single point TDM" In principle, it can not cope with such a complex clinical treatment shared by multiple drugs and the prediction of drug-drug interaction (DDI). In vivo probe is an effective method to evaluate the influence of the body on the attribute law of drugs in vivo. Only based on the effective discrimination of the attribute law of drugs in vivo, can we obtain a complete prediction of the change law of a specific drug, and turn the passive technical method of blood concentration detection into initiative.

DOXO is a metabolism-oriented drug, which is metabolized by CYP1A to TA, which further metabolizes TAA and ETO, so the amount of TAA and ETO can represent the activity of CYP1A, We will explore the method of detecting DOXO kinetics by Vmax method through clinical research. The entire clinical study is divided into two stages, the first stage is the solution of Vmax, and the second stage is the verification of the overall pharmacokinetics. Clinically, multi-drug combination is very easy to produce DDI, and the production of DDI is nothing more than pharmacodynamics or pharmacokinetic interactions. Therefore, when combining drugs or applying acupuncture and drug combination, it is also necessary to monitor the effects and effects of metabolic enzymes in the body on the drugs, and then to determine the safety and the mechanism of the effect of multi-drug sharing. Therefore, further explore acupuncture. Combined with the pharmacokinetic law of DOXO to explore the mechanism of the combined action of acupuncture and medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pneumothorax or three and three lower rib fractures.
2. Age ≥18 years old and ≤40 years old, no gender limit;
3. No chronic underlying disease, no new onset or acute disease;
4. No long-term drug use history;
5. Understand and agree to participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Patients who have received EA treatment in the past;
2. Patients with skin infections in the local meridian points;
3. Patients with upper or lower limb nerve injury;
4. Those who have consumed tea, coffee, chocolate and smoked one week before the start of the test;
5. Those suffering from respiratory diseases, hyperthyroidism, sinus tachycardia, and arrhythmia;
6. Patients with severe heart, lung, liver, and kidney function abnormalities, patients with hypertension, patients with active gastric and duodenal ulcers or patients with co-infection;
7. Those who have participated in or are participating in other clinical trials one month before enrollment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
The concentration of DOXO and metabolites | Within ten minutes after the start of administration
  The concentrations of DOXO and its metabolites TA, TAA and ETO in blood were detected by LC-MS